CLINICAL TRIAL: NCT06553885
Title: A Phase II Study of Enfortumab Vedotin in Patients With Advanced or Metastatic Colorectal Cancer or Hepatocellular Carcinoma
Brief Title: Ph II Study of Enfortumab Vedotin in Patients With Advanced or Metastatic CRC or HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23188
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer; Hepatocellular Carcinoma
Keywords: Nectin-4; Antibody-drug conjugate; Enfortumab; Colorectal; Hepatocellular carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Hepatocellular | interventions — enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Colorectal Cancer (Experimental): Enfortumab vedotin at a dose of 1.25 mg/kg will be administered as an IV infusion over approximately 30 minutes on Days 1, 8, and 15 of every 28-day cycle.
  Interventions: Drug: Enfortumab Vedotin
- Cohort 2: Hepatocellular Carcinoma (Experimental): Enfortumab vedotin at a dose of 1.25 mg/kg will be administered as an IV infusion over approximately 30 minutes on Days 1, 8, and 15 of every 28-day cycle.
  Interventions: Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Enfortumab Vedotin — Enfortumab vedotin is a type of prescription medicine known as an antibody-drug conjugate.
  Other Names: PADCEV

SUMMARY:
This study is a multi-indication, open-label, single-treatment arm, parallel-cohort phase II study of enfortumab vedotin in adult participants with advanced or metastatic colorectal cancer (CRC) or hepatocellular carcinoma (HCC) who have been previously treated with one or more lines of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed CRC or HCC that is metastatic or unresectable and have progressive disease or intolerance after standard front-line therapies as defined below:

Participants with CRC (cohort 1): Participants must have had progressive disease or intolerance after at least 2 but no more than 3 prior lines of systemic therapy in advanced or metastatic setting. Prior lines of therapy should include fluoropyrimidine (5-fluorouracil or capecitabine), oxaliplatin, and irinotecan with or without anti EGFR antibody for RAS/RAF wild-type CRC or bevacizumab unless contraindicated. For patients with microsatellite instability high (MSI-H) CRC, previous lines of therapy should include a PD-1/PD-L1 immune checkpoint inhibitor in additional to the chemotherapy agents mentioned above. Adjuvant chemotherapy with radiographic progression greater than 12 months after the last dose is not considered as a line of therapy.

Participants with HCC (cohort 2): Participants must have had progressive disease or intolerance after at least 1 but no more than 2 prior lines of systemic therapy in advanced or metastatic setting. Prior lines of therapy should include a PD-1/PD-L1 immune checkpoint inhibitor or a multikinase inhibitor, which was administered either alone or in combination.

* Participants must have measurable disease according to RECIST v1.1. Lesions in a prior radiation field must have progressed subsequent to radiotherapy to be considered measurable.
* Participants must have had progression or recurrence of CRC or HCC during or following receipt of most recent therapy.
* Legally an adult according to local regulation at the time of signing informed consent, and minimum age of 18 years
* ECOG performance status ≤1
* Participants must have adequate organ and marrow function as defined below:

  1. Absolute neutrophil count (ANC) ≥ 1500/mm3
  2. Platelet count ≥100 × 109/L
  3. Hemoglobin ≥9 g/dL
  4. Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) or ≤ 3 × ULN for subjects with Gilbert's disease
  5. Creatinine clearance (CrCl) ≥30 mL/min as estimated per institutional standards
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN or ≤ 5 x ULN for subjects with liver metastases
  7. Liver function status should be Child-Pugh (CP) Class A.
* Tumor tissue samples must be available for submission prior to study treatment.
* Participants must have an anticipated life expectancy of ≥3 months as assessed by the investigator.
* The effects of enfortumab vedotin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 4 months after the last dose. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Radiotherapy or major surgery or chemotherapy, biologics, investigational agents, and/or immunotherapy that is not completed 2 weeks prior to first dose of study drug.
* Ongoing sensory or motor neuropathy Grade ≥2. Ongoing clinically significant toxicity (Grade 2 or higher) associated with prior treatment (including systemic therapy, radiotherapy or surgery).
* Active central nervous system (CNS) metastases. Participants with treated CNS metastases are permitted on study if all the following are true: i. CNS metastases have been clinically stable for at least 6 weeks prior to screening and baseline scans show no evidence of new or enlarged metastasis ii. If requiring steroid treatment for CNS metastases, the patient is on a stable dose ≤20 mg/day of prednisone or equivalent for at least 2 weeks iii. Participant does not have leptomeningeal disease
* Prior enrollment in an enfortumab vedotin study or prior treatment with other MMAE-based ADCs.
* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Participants with nonmelanoma skin cancer, localized prostate cancer treated with curative intent with no evidence of progression, low-risk or very low-risk (per standard guidelines) localized prostate cancer under active surveillance/watchful waiting without intent to treat, or carcinoma in situ of any type (if complete resection was performed) are allowed.
* Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of enfortumab vedotin. Routine antimicrobial prophylaxis is permitted.
* Patients with a positive hepatitis B surface antigen and/or antihepatitis B core antibody. Patients with a negative polymerase chain reaction (PCR) assay (HBV DNA is less than 10 IU/ml) are permitted with appropriate antiviral prophylaxis.
* Active hepatitis C infection or known human immunodeficiency virus (HIV) infection. Patients who have been treated for hepatitis C infection are permitted if they have negative HCV RNA test (less than 15 IU/ml) and have documented sustained virologic response of ≥12 weeks.
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of enfortumab vedotin.
* Known hypersensitivity to enfortumab vedotin or to any excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate, and polysorbate 20)
* Participants with active keratitis or corneal ulcerations. Patients with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator.
* Participants with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7-8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained.
* Participants with uncontrolled tumor-related bone pain or impending spinal cord compression, uncontrolled intercurrent illness, psychiatric illness/social situations that would limit compliance with study requirements or other underlying medical condition that, in the opinion of the investigator, would impair the ability of the patient to receive or tolerate the planned treatment and follow-up.
* Pregnant women are excluded from this study because enfortumab vedotin is an antibody-drug conjugate agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with enfortumab vedotin. Breastfeeding should be discontinued if the mother is treated with EV, and for 3 weeks after the last dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 3 years
  The ORR is defined as the proportion of evaluable patients with confirmed CR or PR according to RECIST v1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 3 years
  The DOR is defined as the time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of PD (per RECIST v1.1) or to death due to any cause, whichever comes first.
Progression-free Survival (PFS) | Up to 3 years
  PFS is defined as the time from start of study treatment to first documentation of objective tumor progression (PD per RECIST v1.1), or to death due to any cause, whichever comes first.
Overall Survival (OS) | Up to 3 years
  OS is defined as the time from start of study treatment to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Biachi de Castria, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States